CLINICAL TRIAL: NCT00615966
Title: A Phase 2, Two-Part Study of the Safety and Tolerability of Diannexin in Kidney Transplant Recipients
Brief Title: Phase 2 Study of the Safety of Diannexin in Kidney Transplant Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alavita Pharmaceuticals Inc (Industry)
Collaborators: CTI Clinical Trial and Consulting Services (Other)
Responsible Party: Gordon Ringold, PhD, Alavita Pharmaceuticals Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DAV-CL002
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2011-06-29 (Estimated); Status verified 2011-06

CONDITIONS: Kidney Transplantation
Keywords: kidney transplantation; ischemia-reperfusion injury; phosphatidylserine binding
MeSH Terms: conditions — Reperfusion Injury | interventions — diannexin, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Diannexin
- 2 (Experimental)
  Interventions: Drug: Diannexin
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diannexin — single dose, 200 µg/kg IV
  Arms: 1
Drug: Placebo — Single dose, IV
  Arms: 3
Drug: Diannexin — Single dose, 400 µg/kg IV
  Arms: 2

SUMMARY:
The purpose of this study is evaluate the safety and tolerability of Diannexin in kidney transplant recipients.

DETAILED DESCRIPTION:
Ischemia-reperfusion injury, which occurs when the blood supply to an organ, or part of an organ, is cut off and subsequently restored, is an important clinical problem in the organ transplant setting. Diannexin, a recombinant form of the endogenous human Annexin V protein, is in development as a therapeutic agent designed to prevent ischemia-reperfusion injury following organ transplantation. Pharmacology studies indicate that Diannexin has protective effect in various ischemia-reperfusion injury and organ transplantation models. Diannexin binds to phosphatidylserine on cell surfaces, which is believed to underlie its ability to attenuate ischemia-reperfusion injury. In a completed Phase 1 trial, Diannexin was judged safe and well tolerated in healthy adult subjects. The present study is designed to determine the safety and tolerability of single escalating doses of Diannexin in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive a kidney transplant from a deceased expanded criterion donor (ECD) or a donor cardiac death (DCD) donor that was exposed to no more than 36 hr of cold ischemia prior to transplantation, or scheduled to receive a kidney transplant from a standard criterion donor (SCD) that was exposed to 24-36 hr of cold ischemia prior to transplantation
* Willing to use adequate contraception for at least 4 weeks after dosing
* Willing and able to provide written Informed Consent and to comply with the requirements of the study

Exclusion Criteria:

* If female, subject is pregnant or lactating
* Known bleeding diathesis
* INR at Screening > 1.5
* Platelet count at Screening below LLN and judged clinically significant
* Use of Plavix, anticoagulants other than aspirin, antithrombotics, and/or blood-thinning agents within 10 days prior to study entry
* Previous receipt of an organ transplant
* Will receive concurrent transplant of any additional organ(s)
* Clinically significant active infection at study entry
* Surgery within 2 weeks prior to study entry
* Believed to have used an illicit drug and/or abused alcohol within 3 months prior to study entry
* Presence of a psychiatric illness that might interfere with study participation
* Cancer, other than basal cell or squamous cell cancer of the skin, within 2 years prior to study entry
* Scheduled to receive a kidney transplant from a low risk donor
* Currently participation, or participated within 30 days prior to study entry, in an investigational drug study
* Known allergy to kanamycin
* History or presence of any medical condition or disease that could place the subject an unacceptable risk for study participation

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Safety assessments -- physical examinations, vital signs, clinical safety laboratory tests, ECGs, immunogenicity testing, adverse events | 28 days following administration of study medication

SECONDARY OUTCOMES:
Population pharmacokinetics | Through Hour 48 after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Knechtle, MD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - University of Maryland, Baltimore, Maryland
  - St Barnabas Medical Center, Livingston, New Jersey
  - New York-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - University of Wisconsin Medical School, Dept of Surgery, Madison, Wisconsin

REFERENCES:
- [Derived] Cheng EY, Sharma VK, Chang C, Ding R, Allison AC, Leeser DB, Suthanthiran M, Yang H. Diannexin decreases inflammatory cell infiltration into the islet graft, reduces beta-cell apoptosis, and improves early graft function. Transplantation. 2010 Oct 15;90(7):709-16. doi: 10.1097/TP.0b013e3181ed55d8. PMID 20634785